CLINICAL TRIAL: NCT00122291
Title: A Phase 2 Study of Preoperative Radiation Therapy and Capecitabine (an Oral Fluoropyrimidine Carbamate) in Locally Advanced Rectal Cancer
Brief Title: A Study of Preoperative Radiation Therapy and Capecitabine in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16080; Capecitabine Phase 2
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2011-08

CONDITIONS: Rectal Cancer; Neoplasm Metastasis
Keywords: preoperative; chemotherapy; radiation therapy; rectal cancer; transmural rectal wall invasion; nodal metastasis
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis | interventions — Capecitabine

INTERVENTIONS:
Drug: Capecitabine
Procedure: Pelvic radiation

SUMMARY:
The purpose of this trial is to study the efficacy of preoperative radiation therapy and capecitabine in locally advanced rectal cancer.

DETAILED DESCRIPTION:
The purpose of this trial is to study the efficacy of preoperative radiation therapy and capecitabine in locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy - proven rectal cancer
* Transmural rectal wall invasion
* Karnofsky performance status >70
* Normal bone marrow, liver and kidney function

Exclusion Criteria:

* Distant metastases
* Prior pelvic radiation
* Inflammatory bowel disease
* Severe ischemic heart disease
* Anticoagulant therapy
* Pregnancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2002-01

PRIMARY OUTCOMES:
safety
response

CONTACTS AND LOCATIONS:
Overall Officials: Gwyn Bebb, MD, Principal Investigator — Alberta Health services
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada